CLINICAL TRIAL: NCT02732743
Title: An Open Label, Non-comparative Pilot Study to Assess the Efficacy and Safety of the Food Supplement Physiomanna® Baby in Pediatric Patients With a History of Functional Constipation
Brief Title: Food Supplement Physiomanna® Baby in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuppa Industriale Srl (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IU01/016
Record Dates: First submitted 2016-03-31; First posted 2016-04-11 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2017-03

CONDITIONS: Irritable Bowel Syndrome Characterized by Constipation
Keywords: childhod constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Food Supplement Physiomanna® Baby (Other): Dosage: 1g/kg body
  Interventions: Dietary Supplement: Physiomanna® Baby

INTERVENTIONS:
Dietary Supplement: Physiomanna® Baby — Dosage 1g/kg body, 2 cycles (if applicable)

SUMMARY:
The primary objective is to assess the efficacy and safety of the Food Supplement Physiomanna® Baby in pediatric patients with a history of functional constipation

The secondary objective of the trial is to evaluate the adherence to product's administration in the enrolled children.

DETAILED DESCRIPTION:
This is an interventional, non-controlled, multicenter trial with a prospective design in one cohort of patients. This clinical investigation will be performed in 3 centers in Romania.

The tested hypothesis is that Physiomanna® Baby administration for 3 weeks, increases the SBM to be more than 2 times per week.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients between the ages of 0 to 8 years;
* Functional constipation according to ROME III criteria (Annex 2);
* Two or fewer SBM during the previous week; SBM is defined as BM not preceded after a 24 h administration with a laxative or enema;
* To be otherwise in good health, as judged by a physical examination;
* Mentally competent parent or tutor to sign an informed consent

Exclusion Criteria:

* Known history of organic cause for the constipation;
* Congenital malformations that produce constipation (Hirschsprung's disease, imperforate anus, children with cerebral palsy or other neurologic abnormalities, or systemic diseases);
* Fecal Occult Blood Test (FOBT) positive in the 4 previous weeks;
* Fecal impaction at baseline, or during the trial period, as indicated by the physical examination;
* Known or suspected perforation or obstruction other than fecal impaction;
* History of gastric retention, inflammatory bowel disease, bowel resection, or colostomy;
* Use of concomitant medications that cause constipation in the previous 3 months;
* Concomitant use of herbs and other dietary supplements, such as: stimulant laxative herbs and/or potassium depleting herbs;
* Concomitant use of cardiac glycosides(e.g. Digoxin);
* Patients who, according to the investigator, should not be included in the study for any reason, including the parent's inability to follow the study procedures;
* Patients with known allergy to Fraxinus Manna, mannitole, fennel, lemon balm or chamomile;
* Patients with clinically significant elevations of TSH or abnormal plasma electrolytes in the 4 previous weeks;
* Patients who, within the past 30 days have participated in an investigational clinical study;

Ages: 1 Week to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of Spontaneous Bowel Movements (SBM) per week | 2-3 weeks

SECONDARY OUTCOMES:
Safety: Adverse Events (AE) check; Investigator and Patient Global Assessment | 2-3 weeks

OTHER OUTCOMES:
Investigator and Patient Global Assessment for Efficacy | 2-3 weeks
Analysis of product's administration adherence by diary cards | 2-3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barattini Dionisio, MD, Study Director — Opera CRO
Locations (1):
- Opera Contract Research Organization SRL, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tabbers MM, Boluyt N, Berger MY, Benninga MA. Clinical practice : diagnosis and treatment of functional constipation. Eur J Pediatr. 2011 Aug;170(8):955-63. doi: 10.1007/s00431-011-1515-5. Epub 2011 Jun 24. PMID 21701812
- [Background] Tabbers MM, Boluyt N, Berger MY, Benninga MA. Nonpharmacologic treatments for childhood constipation: systematic review. Pediatrics. 2011 Oct;128(4):753-61. doi: 10.1542/peds.2011-0179. Epub 2011 Sep 26. PMID 21949142
- [Background] Loening-Baucke V, Miele E, Staiano A. Fiber (glucomannan) is beneficial in the treatment of childhood constipation. Pediatrics. 2004 Mar;113(3 Pt 1):e259-64. doi: 10.1542/peds.113.3.e259. PMID 14993586
- [Background] Livesey G. Health potential of polyols as sugar replacers, with emphasis on low glycaemic properties. Nutr Res Rev. 2003 Dec;16(2):163-91. doi: 10.1079/NRR200371. PMID 19087388
- [Background] Caligiani A, Tonelli L, Palla G, Marseglia A, Rossi D, Bruni R. Looking beyond sugars: phytochemical profiling and standardization of manna exudates from Sicilian Fraxinus excelsior L. Fitoterapia. 2013 Oct;90:65-72. doi: 10.1016/j.fitote.2013.07.002. Epub 2013 Jul 10. PMID 23850543
- [Background] Kountouras J, Magoula I, Tsapas G, Liatsis I. The effect of mannitol and secretin on the biliary transport of urate in humans. Hepatology. 1996 Feb;23(2):229-33. doi: 10.1053/jhep.1996.v23.pm0008591845.
- [Background] Taylor SN, Basile LA, Ebeling M, Wagner CL. Intestinal permeability in preterm infants by feeding type: mother's milk versus formula. Breastfeed Med. 2009 Mar;4(1):11-5. doi: 10.1089/bfm.2008.0114. PMID 19196035